CLINICAL TRIAL: NCT02137044
Title: Improving the Quality of Care for Pain and Depression in Persons With Multiple Sclerosis
Brief Title: Multiple Sclerosis-Collaborative Approach to Rehabilitation Effectiveness Study
Acronym: MS-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Dawn Ehde, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46597; 46597 (Other: UW IRB)
Record Dates: First submitted 2014-04-22; First posted 2014-05-13 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Multiple Sclerosis; Pain; Depression
Keywords: multiple sclerosis; pain; depression
MeSH Terms: conditions — Multiple Sclerosis; Pain; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Care (CC) (Experimental): Collaborative care (CC) is a systematic and integrated approach to improving the delivery and utilization of effective treatments for chronic pain and depression. The care was delivered through an interdisciplinary team, organized around a CC manager (CCM) who guided the patient through various aspects of care during the 16-week treatment phase. The team also included the patient's MS physician and the CC Supervisors, a group of clinicians who were experts of the study domain . The CCM offered all subjects care management, collaborative medical management, and psychosocial treatment appropriate to their problem area (i.e., pain, depression, or both) described below. If the patient had both pain and depression, he or she received care management and collaborative medical management for both.
  Interventions: Behavioral: Collaborative Care (CC)
- Usual Care (No Intervention): Subjects assigned to usual care were informed by the CCM of their depressive and pain symptoms and that they should consult with their MS or primary care provider about possible care for these conditions. Study personnel did not make any further attempts to influence usual care participants' depression or pain management unless a psychiatric emergency arose (e.g., suicidal ideation was detected at baseline or any of the outcome assessments).

INTERVENTIONS:
Behavioral: Collaborative Care (CC) — Collaborative care (CC) is a systematic and integrated approach to improving the delivery and utilization of effective treatments for chronic pain and depression. The care was delivered through an interdisciplinary team, organized around a CC manager (CCM) who guided the patient through various aspects of care during the 16-week treatment phase. The team also included the patient's MS physician and the CC Supervisors, a group of clinicians who were experts of the study domain . The CCM offered all subjects care management, collaborative medical management, and psychosocial treatment appropriate to their problem area (i.e., pain, depression, or both) described below. If the patient had both pain and depression, he or she received care management and collaborative medical management for both.
  Arms: Collaborative Care (CC)

SUMMARY:
The purpose of this study is to: (1) test the benefits of the patient-centered collaborative care treatment approach for persons with MS who also have depression and/or pain; and also (2) test whether this approach improves quality of life, patient satisfaction, adherence to other treatments, and quality of care in the MS care system.

DETAILED DESCRIPTION:
Background: It is common for people with multiple sclerosis (MS) to have depression and chronic pain. Individuals with MS who have depression and/or pain often use more health care services, benefit less from treatment, and have poorer quality of life. While evidence-based medical and behavioral treatments for depression and pain exist, they are often not offered or accessible to persons with MS. As a result, chronic pain and depression are under-treated in people with MS. One way to better treat these problems is through a "Collaborative Care" approach. In this approach a care manager (nurse supervised by expert physicians, psychiatrists, and psychologists) helps coordinate and provide high-quality, evidence-based treatments for depression and pain. The care manager also makes sure that the care is focused on the patient's goals and preferences. The care is provided by phone or in person based on the patient's preference. Although this approach has been used successfully with patients with many different conditions, it has never been tested in patients with MS, pain, and depression.

Objectives: The investigators' objectives are to (1) test the benefits of the patient-centered collaborative care treatment approach for persons with MS who also have depression and/or pain; and also (2) test whether this approach improves quality of life, patient satisfaction, adherence to other treatments, and quality of care in the MS care system.

Methods: Participants were 195 outpatients with MS from a specialty MS Center who had depression and/or chronic pain. Half of the participants received the treatment that was typical for patients in the MS Center ("usual care"), while the other half received treatment using the Collaborative Care approach. Participants in the collaborative care group met regularly in-person or by telephone with a social worker who coordinated their depression and pain treatments and provided strategies for better managing their symptoms. The treatment phase of the study lasted for 16 weeks and began within 2 weeks of study enrollment. Participants completed telephone interviews within 2 weeks of enrollment, approximately 4 months after study enrollment, and approximately 10 months after study enrollment. During these interviews participants were asked questions about their pain, depression, satisfaction with care, and quality of life to compare the two care approaches.

Projected Patient Outcomes: The investigators anticipate that those in the collaborative care approach will have better controlled pain and depression and better quality of life, satisfaction with care, adherence to other MS treatments, and quality of care compared to those in the usual care approach. The results of this study may help patients, clinicians, healthcare system leaders, and policy makers make decisions about the benefits of this type of coordinated care approach for depression and pain in MS care.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a definitive diagnosis of MS confirmed by subjects' MS physician in the University of Washington (UW) MS Center;
* Patient has received care and plans to continue to receive care at the UW MS Center during enrollment period;
* Patient has access to and is able to communicate over the telephone (we will provide phone headsets if needed) to allow participation in the telehealth components of the study;
* Patient can read, speak and understand English;
* Patient is at least 18 years of age.
* Patient reports a clinically significant problem with pain and/or depression.

Exclusion Criteria:

* Patient represents a high suicide risk;
* Patient reports symptoms of a current psychotic disorder or diagnosis of bipolar disorder with current psychotic features at time of screening;
* Subject attends appointments more than once per month with a psychiatrist for treatment of depression;
* Patient reports planning major surgery in the next ten months;
* Patient reports alcohol or psycho-active substance dependence within past month;
* Patient has moderate to severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in Control of Pain | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  Control of pain is defined as either average pain severity score of less than 3 in the past week on the Brief Pain Inventory, or obtaining a 30% or greater reduction in average pain severity from baseline. Pain severity will be assessed using the Brief Pain Inventory 0-10 numerical rating scale.
Change in Control Of Depression | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  Control of depression is defined as a reduction of at least 50% depression severity or a score of < 0.5 on the SCL-20. Depression severity will be assessed with the Symptom Checklist Depression Subscale (SCL-20), a brief self-report measure of cognitive, emotional and somatic symptoms of depression commonly used in treatment outcome studies.

SECONDARY OUTCOMES:
Change in Depression Severity | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  Depression severity, as measured by the SCL-20, will be assessed as a continuous measure of depression symptom severity.
Change in Quality of Depression Care | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  The investigators will assess the proportion of participants who achieve guideline-level depression care. For depression this is defined as: use of antidepressant at therapeutic dose 25 of the past 30 days, or at least 4 evidence-based psychotherapy sessions since the last assessment period (or 6 months, whichever is shorter). The investigators will also determine whether participants have a diagnosis of major depressive disorder or dysthymia using modules from the Mini International Neuropsychiatric Interview (MINI), which will be administered by telephone by trained staff.
Change in Pain Severity | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  Pain severity, as measured by the Brief Pain Inventory 0-10 NRS scale, will be assessed as a continuous measure of pain severity.
Change in Disability | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  The investigators will use the Sheehan Disability Scale, a 3-item measure that assesses how diminished health status interferes with work/school, family life, and social life and activities.
Change in Health-Related Quality of Life | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  The investigators will administer the EuroQol EQ-5D, a standardized measure of health status. It is comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Improvement and Satisfaction with Care | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  The investigators will use the Patient Global Impression of Change scale, a single question which asks participants to rate their improvement with treatment on a 7-point scale that ranges from "very much improved" to "very much worse," with "no change" as the mid-point. In addition, a single question will be used to ask participants to rate their overall satisfaction with their care on a 0 to 4 scale that ranges from "very dissatisfied" to "very satisfied."

OTHER OUTCOMES:
Change in Fatigue | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  Given the potential for fatigue to improve should pain and/or depression improve, the investigators will administer the PROMIS Fatigue-MS (Short-Form) to assess the effects, if any, of the intervention on fatigue.
Change in Healthcare Utilization | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  The Cornell Service Index is a widely used measure of healthcare services utilization, and will include number of hospitalizations and days hospitalized, number of emergency department visits, as well as clinic visits (both routine and those that address medical complications).
Change in Self-Efficacy | Within 2 weeks following study enrollment, about 4 Months following study enrollment, about 10 months following study enrollment
  Self-efficacy is hypothesized to be an important determinant of self-management in chronic diseases, including MS. The PROMIS MS-self-efficacy scale, which has strong psychometric properties, will be used to determine if patients' perceived self-efficacy specific to managing MS changes as a result of the collaborative care intervention.
Change in Pain Severity | During each treatment session for subjects randomized to collaborative care intervention assignment. These subjects will participate in 10-12 treatment sessions over a 16-week period that starts about 1-2 weeks after study enrollment.
  Numerical Rating Scale-11 (NRS-11): Average pain intensity over the past week will be assessed using an 11-point NRS.
Change in Depression Severity | During each treatment session for subjects randomized to collaborative care intervention assignment. These subjects will participate in 10-12 treatment sessions over a 16-week period that starts about 1-2 weeks after study enrollment.
  Patient Health Questionnaire-9 (PHQ-9) is a nine item measure of depression symptoms that parallels the DSM-IV criteria for major depression. A score of 10 or more has high sensitivity and specificity for major depression.
Descriptive Characteristics | Within 2 weeks of enrollment
  Descriptives will be collected at baseline from the medical record and patient self-report. They will include demographic variables (sex, age, race, ethnicity, education level, employment status, postal zip code, and marital status) and MS variables [date of MS diagnosis, course of MS -relapsing-remitting, primary-progressive, secondary-progressive, or progressive-relapsing, current Expanded Disability Status Scale(EDSS) score (a core measure of MS disease progression in clinical trials),and use of disease-modifying medications]. We will also collect information describing participants' pain and depression histories, including pain sites, number of pain sites, pain duration, and depression history.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Ehde, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of Washington- Harborview Medical Center, Seattle, Washington
  - University of Washington Medicine MS Center, Seattle, Washington
  - University of Washington-Health Sciences Building, Seattle, Washington

REFERENCES:
- [Derived] Ehde DM, Alschuler KN, Sullivan MD, Molton IP, Ciol MA, Bombardier CH, Curran MC, Gertz KJ, Wundes A, Fann JR. Improving the quality of depression and pain care in multiple sclerosis using collaborative care: The MS-care trial protocol. Contemp Clin Trials. 2018 Jan;64:219-229. doi: 10.1016/j.cct.2017.10.001. Epub 2017 Oct 5. PMID 28987615